CLINICAL TRIAL: NCT00307034
Title: An Open, Randomized, Phase IIIa Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine, When Administered Intramuscularly According to a 2-4-11 Months Vaccination Schedule
Brief Title: Safety & Immunogenicity Study of 10-Valent Pneumococcal Conjugate Vaccine When Administered as a 2-Dose Schedule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 105539
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2017-02

CONDITIONS: Infections, Streptococcal
Keywords: Primary vaccination; Pneumococcal disease; Safety; Booster vaccination; Immunogenicity; Pneumococcal vaccine; Dose comparison
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (2):
- 2-dose group (Experimental): Subjects receiving GSK Biologicals' 10-valent pneumococcal conjugate vaccine at 2-4-11 months of age, co-administered with DTPa-combined vaccine (Infanrix hexa or Infanrix IPV/Hib) at 2-4-11 months of age.
  Interventions: Biological: GSK Biologicals' 10-valent pneumococcal conjugate vaccine.; Biological: Infanrix hexa.; Biological: Infanrix-IPV/Hib.
- Comparator group (Experimental): Subjects receiving GSK Biologicals' 10-valent pneumococcal conjugate vaccine at 2-3-4-11 months of age, co-administered with DTPa-combined vaccine (Infanrix hexa or Infanrix IPV/Hib) at 2-4-11 months of age.
  Interventions: Biological: GSK Biologicals' 10-valent pneumococcal conjugate vaccine.; Biological: Infanrix hexa.; Biological: Infanrix-IPV/Hib.

INTERVENTIONS:
Biological: GSK Biologicals' 10-valent pneumococcal conjugate vaccine. — Intramuscular injection, 3 or 4 doses (2-4-11 or 2-3-4-11 months of age schedule).
Biological: Infanrix hexa. — Intramuscular injection, 3 doses (2-4-11 months of age schedule).
  Other Names: DTPa-HBV-IPV/Hib
Biological: Infanrix-IPV/Hib. — Intramuscular injection, 3 doses (2-4-11 months of age schedule).
  Other Names: DTPa-IPV/Hib

SUMMARY:
Assess immuno, reacto of the 10-valent pneumococcal vaccine after 2 doses (2, 4 months of age) and after the complete 2, 4, 11 months schedule when co-administered with DTPa-HBV-IPV/Hib or DTPa-IPV/Hib (according to national recommendations)

DETAILED DESCRIPTION:
Total anticipated: 300 subjects (150/group). 2-dose group - 10-valent pneumococcal vaccine + DTPa combined vaccine (2, 4, 11 months); Comparator group - 10-valent pneumococcal vaccine (2, 3, 4, 11 months) + DTPa combined vaccine (2, 4, 11 months). The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion criteria:

* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 8 and 16 weeks (56-120 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks.

Exclusion criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting 30 days before the first dose of vaccine(s) and ending 30 days after the last dose, with exception of BCG vaccination which can be given after the 1 month post-dose 2 or 3 (2-4-11 or 2-3-4-11 months of age schedule) blood sampling and a minimum of 30 days before the pre-booster dose blood sampling.
* Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b, and/or S. pneumoniae.
* History of or intercurrent diphtheria, tetanus, pertussis, hepatitis B, polio, Haemophilus influenzae type b disease, and/or invasive pneumococcal diseases.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 8 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 351 (Actual)
Dates: Start 2006-01-01; Primary Completion 2007-01-01 (Actual); Study Completion 2007-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- GSK Investigational Site, Hvidovre, Denmark
- Norway (2):
  - GSK Investigational Site, Morvik
  - GSK Investigational Site, Oslo
- Slovakia (2):
  - GSK Investigational Site, Dolný Kubín
  - GSK Investigational Site, Ružomberok
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Umeå

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Schuerman L et al. Population variability in antibody responses following pneumococcal conjugate vaccination: experience with the non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. Population variability of opsonophagocytic activity following 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate (PHiD-CV) vaccination more limited than antibody responses. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. Prevention of invasive pneumococcal disease and meningitis with PHiD-CV when used according to a 2+1 schedule. Abstract presented at the Meningitis Research Foundation Conference (MRFC). London, UK, 11-12 November 2009.
- [Background] Silfverdal SA, Hogh B, Bergsaker MR, Skerlikova H, Lommel P, Borys D, Schuerman L. Immunogenicity of a 2-dose priming and booster vaccination with the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine. Pediatr Infect Dis J. 2009 Oct;28(10):e276-82. doi: 10.1097/INF.0b013e3181b48ca3. PMID 20118683
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 105539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105539 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Synflorix I Group: Healthy male or female subjects between and including 8 to 16 weeks (56-120 days) of age at the time of first vaccination, received a 2-dose primary vaccination course of Synflorix™ (10Pn-PD-DiT) vaccine at 2 and 4 months of age, followed by a booster dose of the same vaccine at 11 months of age, each dose being co-administered with one dose of Infanrix Hexa™ (DTPa-HBV-IPV/Hib) or Infanrix™-IPV/Hib (DTPa-IPV/Hib), according to national recommendations. Synflorix™ vaccine was administered intramuscularly into the right antero-lateral thigh and Infanrix™ combined vaccine was administered intramuscularly into the left antero-lateral thigh.
- Synflorix II Group: Healthy male or female subjects between and including 8 to 16 weeks (56-120 days) of age at the time of first vaccination, received a 3-dose primary vaccination course of Synflorix™ (10Pn-PD-DiT) vaccine at 2, 3 and 4 months of age, co-administered with 2 doses of Infanrix Hexa™ (DTPa-HBV-IPV/Hib) or Infanrix™-IPV/Hib (DTPa-IPV/Hib) at 2 and 4 months of age, followed by a booster dose of the Synflorix™ vaccine at 11 months of age, co-administered with one dose of the Infanrix™ combined vaccine, according to national recommendations. Synflorix™ vaccine was administered intramuscularly into the right antero-lateral thigh and Infanrix™ combined vaccine was administered intramuscularly into the left antero-lateral thigh.
Period: Overall Study
Arm/Group | Synflorix I Group | Synflorix II Group
Started | 175 | 176
Completed | 173 | 169
Not Completed | 2 | 7
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix I Group | Synflorix II Group | Total
Number analyzed (Participants) | 175 | 176 | 351
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 12 (1.94) | 12.1 (1.9) | 12.05 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 82 | 168
  Male | 89 | 94 | 183

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Pneumococcal Serotypes
Description: A seroprotected subject was defined as a subject who had anti-pneumococcal serotypes antibody concentrations greater than or equal to (≥) the threshold value of 0.20 micrograms per milliliter (μg/mL). The vaccine pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C,19F and 23F (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs). The results presented for the Group 1 correspond to the primary outcome.
Time Frame: One month post-dose 2 (Month 3) administration of Synflorix™ vaccine
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity concerning data were available.
Measure: Number; unit: Subjects
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 153 | 153
Subjects
  Anti-1 (N= 153, 151) | 149 | 149
  Anti-4 (N=153, 153) | 150 | 152
  Anti-5 (N=152, 149) | 146 | 149
  Anti-6B (N=149, 149) | 83 | 94
  Anti-7F (N=153, 152) | 148 | 151
  Anti-9V (N=152, 153) | 142 | 152
  Anti-14 (N=152, 152) | 146 | 152
  Anti-18C (N=152, 153) | 146 | 152
  Anti-19F (N=152, 152) | 141 | 146
  Anti-23F (N=153, 152) | 106 | 118

2. Secondary Outcome: Number of Seroprotected Subjects Against Pneumococcal Serotypes
Description: A seroprotected subject was defined as a subject who had anti-pneumococcal serotypes antibody concentrations greater than or equal to (≥) the threshold value of 0.20 micrograms per milliliter (μg/mL). The vaccine pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C,19F and 23F (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs).
Time Frame: One month before (Month 9) and one month after (Month 10) the booster dose of Synflorix™ vaccine
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity concerning data were available.
Measure: Number; unit: Subjects
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 156 | 149
Subjects
  Anti-1, Month 9 (N= 149, 147) | 77 | 101
  Anti-1, Month 10 (N=156, 147) | 155 | 147
  Anti-4, Month 9 (N= 152, 149) | 120 | 137
  Anti-4, Month 10 (N=155, 147) | 155 | 147
  Anti-5, Month 9 (N= 148, 149) | 121 | 133
  Anti-5, Month 10 (N=155, 147) | 155 | 147
  Anti-6B, Month 9 (N= 154, 148) | 101 | 111
  Anti-6B, Month 10 (N=156, 147) | 138 | 142
  Anti-7F, Month 9 (N= 151, 149) | 135 | 146
  Anti-7F, Month 10 (N=156, 147) | 156 | 147
  Anti-9V, Month 9 (N= 153, 149) | 133 | 142
  Anti-9V, Month 10 (N=156, 147) | 155 | 147
  Anti-14, Month 9 (N= 151, 149) | 140 | 147
  Anti-14, Month 10 (N=156, 147) | 155 | 145
  Anti-18C, Month 9 (N= 154, 149) | 133 | 144
  Anti-18C, Month 10 (N=156, 147) | 156 | 146
  Anti-19F, Month 9 (N= 153, 149) | 140 | 143
  Anti-19F, Month 10 (N=156, 147) | 150 | 144
  Anti-23F, Month 9 (N= 151, 148) | 108 | 116
  Anti-23F, Month 10 (N=154, 147) | 148 | 141

3. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes
Description: The vaccine pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C,19F and 23F (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (μg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 μg/mL. This outcome concerns results for the Primary and Booster Phases of the study.
Time Frame: One month post-dose 2 or post-dose 3 (Month 3) administration, one month before (Month 9) and one month after (Month 10) the booster dose of Synflorix™ vaccine
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 156 | 153
μg/mL
  Anti-1, Month 3 (N= 153, 151) | 1.03 [0.9 to 1.18] | 1.23 [1.07 to 1.42]
  Anti-1, Month 9 (N= 149, 147) | 0.21 [0.19 to 0.24] | 0.3 [0.26 to 0.34]
  Anti-1, Month 10 (N=156, 147) | 1.85 [1.59 to 2.15] | 1.88 [1.62 to 2.17]
  Anti-4, Month 3 (N= 153, 153) | 1.37 [1.21 to 1.55] | 1.71 [1.47 to 1.99]
  Anti-4, Month 9 (N= 152, 149) | 0.4 [0.35 to 0.46] | 0.64 [0.56 to 0.73]
  Anti-4, Month 10 (N=155, 147) | 3.06 [2.68 to 3.49] | 3.47 [3.03 to 3.98]
  Anti-5, Month 3 (N= 152, 149) | 1.32 [1.14 to 1.52] | 1.85 [1.63 to 2.1]
  Anti-5, Month 9 (N= 148, 149) | 0.43 [0.37 to 0.5] | 0.59 [0.51 to 0.68]
  Anti-5, Month 10 (N=155, 147) | 2.65 [2.31 to 3.03] | 3.21 [2.81 to 3.67]
  Anti-6B, Month 3 (N= 149, 149) | 0.19 [0.15 to 0.24] | 0.31 [0.25 to 0.38]
  Anti-6B, Month 9 (N= 154, 148) | 0.28 [0.23 to 0.35] | 0.44 [0.36 to 0.54]
  Anti-6B, Month 10 (N=156, 147) | 1.12 [0.88 to 1.41] | 1.85 [1.54 to 2.22]
  Anti-7F, Month 3 (N= 153, 152) | 1.28 [1.13 to 1.46] | 2.14 [1.9 to 2.4]
  Anti-7F, Month 9 (N= 151, 149) | 0.55 [0.49 to 0.63] | 0.92 [0.81 to 1.05]
  Anti-7F, Month 10 (N=156, 147) | 2.81 [2.51 to 3.15] | 3.88 [3.45 to 4.37]
  Anti-9V, Month 3 (N= 152, 153) | 0.92 [0.81 to 1.05] | 1.47 [1.29 to 1.68]
  Anti-9V, Month 9 (N= 153, 149) | 0.52 [0.46 to 0.6] | 0.87 [0.77 to 0.99]
  Anti-9V, Month 10 (N=156, 147) | 2.95 [2.59 to 3.37] | 3.97 [3.49 to 4.5]
  Anti-14, Month 3 (N= 152, 152) | 1.72 [1.45 to 2.05] | 2.57 [2.22 to 2.97]
  Anti-14, Month 9 (N= 151, 149) | 0.77 [0.64 to 0.93] | 1.53 [1.27 to 1.85]
  Anti-14, Month 10 (N=156, 147) | 4.19 [3.62 to 4.85] | 5.47 [4.68 to 6.4]
  Anti-18C, Month 3 (N= 152, 153) | 1.26 [1.06 to 1.51] | 3.42 [2.87 to 4.07]
  Anti-18C, Month 9 (N= 154, 149) | 0.59 [0.5 to 0.69] | 1.14 [0.96 to 1.35]
  Anti-18C, Month 10 (N=156, 147) | 6.24 [5.43 to 7.18] | 7.2 [6.08 to 8.52]
  Anti-19F, Month 3 (N= 152, 152) | 2.43 [1.97 to 2.98] | 4.43 [3.6 to 5.45]
  Anti-19F, Month 9 (N= 153, 149) | 1.04 [0.87 to 1.25] | 1.7 [1.41 to 2.04]
  Anti-19F, Month 10 (N=156, 147) | 5.58 [4.65 to 6.69] | 6.95 [5.92 to 8.17]
  Anti-23F, Month 3 (N= 153, 152) | 0.38 [0.3 to 0.47] | 0.52 [0.42 to 0.63]
  Anti-23F, Month 9 (N= 151, 148) | 0.32 [0.26 to 0.4] | 0.44 [0.36 to 0.54]
  Anti-23F, Month 10 (N=154, 147) | 2.41 [1.98 to 2.94] | 2.78 [2.31 to 3.35]

4. Secondary Outcome: Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes
Description: Seropositivity status was defined as the opsonophacocytic activity against pneumococcal serotypes greater than or egual to (≥) the value of 8. The vaccine pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C,19F and 23F (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F).This outcome concerns results for the Primary and Booster Phases of the study.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 136 | 135
Titers
  Opsono-1, Month 3 (N= 130, 132) | 21.9 [16.4 to 29.1] | 26.5 [19.8 to 35.4]
  Opsono-1, Month 9 (N= 136, 134) | 5.1 [4.5 to 5.8] | 6.7 [5.4 to 8.3]
  Opsono-1, Month 10 (N=131, 126) | 109.9 [76.1 to 158.7] | 100.6 [68.9 to 146.9]
  Opsono-4, Month 3 (N= 134, 132) | 462.6 [410.4 to 521.4] | 758.9 [647.8 to 888.9]
  Opsono-4, Month 9 (N= 104, 114) | 13.8 [9.7 to 19.6] | 18.6 [12.7 to 27.2]
  Opsono-4, Month 10 (N=125, 101) | 634.6 [496.3 to 811.3] | 1204 [990.7 to 1463.2]
  Opsono-5, Month 3 (N= 132, 130) | 48.3 [37.7 to 61.8] | 68.4 [54 to 86.5]
  Opsono-5, Month 9 (N= 133, 135) | 9.9 [8.1 to 12] | 10.7 [8.6 to 13.4]
  Opsono-5, Month 10 (N=133, 121) | 102.1 [75.8 to 137.6] | 157.2 [123.1 to 200.7]
  Opsono-6B, Month 3 (N= 125, 126) | 157.8 [104.7 to 237.8] | 379.6 [272.4 to 529.1]
  Opsono-6B, Month 9 (N= 121, 124) | 56.1 [34.9 to 90.4] | 62.9 [40.2 to 98.5]
  Opsono-6B, Month 10 (N=132, 103) | 220.3 [146.9 to 330.3] | 468.5 [311.6 to 704.3]
  Opsono-7F, Month 3 (N= 127, 131) | 844.8 [591.4 to 1206.7] | 2176.5 [1759.2 to 2692.7]
  Opsono-7F, Month 9 (N= 113, 126) | 148.5 [89.5 to 246.4] | 380.6 [253 to 572.6]
  Opsono-7F, Month 10 (N=128, 109) | 1843.4 [1494.2 to 2274.1] | 3290.6 [2709.1 to 3996.8]
  Opsono-9V, Month 3 (N= 134, 132) | 875.1 [732 to 1046.1] | 1343.4 [1130.8 to 1596]
  Opsono-9V, Month 9 (N= 120, 134) | 266.8 [205.1 to 347.1] | 322.2 [256.4 to 405.1]
  Opsono-9V, Month 10 (N=129, 109) | 1068.1 [874.7 to 1304.2] | 1706.9 [1438.5 to 2025.3]
  Opsono-14, Month 3 (N= 132, 131) | 692.6 [559.1 to 858] | 1125.3 [946.2 to 1338.3]
  Opsono-14, Month 9 (N= 102, 123) | 52.1 [32.4 to 84] | 157.3 [108.5 to 228.1]
  Opsono-14, Month 10 (N=107, 101) | 835.5 [672.1 to 1038.5] | 1280.7 [1054.5 to 1555.5]
  Opsono-18C, Month 3 (N= 134, 131) | 56.2 [42.9 to 73.7] | 218.6 [176.1 to 271.4]
  Opsono-18C, Month 9 (N= 122, 126) | 8.3 [6.5 to 10.7] | 16.9 [12.5 to 22.8]
  Opsono-18C, Month 10 (N=136, 130) | 330 [259.1 to 420.3] | 490.8 [395.3 to 609.4]
  Opsono-19F, Month 3 (N= 131, 128) | 101 [74.9 to 136] | 356.7 [263.2 to 483.4]
  Opsono-19F, Month 9 (N= 130, 134) | 16.5 [12.9 to 21.1] | 31.6 [24.5 to 40.8]
  Opsono-19F, Month 10 (N=131, 129) | 251.3 [193.4 to 326.6] | 734.7 [568.3 to 949.8]
  Opsono-23F, Month 3 (N= 131, 129) | 489.7 [342.6 to 700] | 1233.7 [991.7 to 1534.7]
  Opsono-23F, Month 9 (N= 112, 133) | 190.7 [115.2 to 315.6] | 150.7 [95.9 to 236.8]
  Opsono-23F, Month 10 (N=134, 121) | 1047.3 [748.1 to 1466.3] | 1528.9 [1171.2 to 1996]

5. Secondary Outcome: Antibody Concentrations Against Protein D (Anti-PD)
Description: Anti-protein D concentrations are expressed as geometric mean concentrations (GMCs), in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).Seropositivity status was defined as Anti-PD antibody concentrations greater than or equal to (≥) the value of 100 EL.U/mL. This outcome concerns results for the Primary and Booster Phases of the study.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 154 | 148
EL.U/mL
  Anti-PD, Month 3 (N=149, 148) | 861.8 [740.4 to 1003.1] | 1223.3 [1066.5 to 1403.2]
  Anti-PD, Month 9 (N= 151, 148) | 349.7 [294.2 to 415.7] | 499.8 [425.3 to 587.2]
  Anti-PD, Month 10 (N= 154, 146) | 1629.8 [1346.4 to 1972.8] | 2113 [1808.9 to 2468.2]

6. Secondary Outcome: Antibody Concentrations Against Diphteria (Anti-D) and Tetanus (Anti-T) Toxoids
Description: Concentrations of antibodies are presented as geometric mean concentrations, expressed as international units per milliliter (IU/mL). Seroprotection status was defined as anti-diphteria and anti-tetanus toxoid antibody concentrations greater than or equal to (≥) the value of 0.1 IU/mL. This outcome concerns results for the Primary and Booster Phases of the study.
Time Frame: One month post-dose 2 (Month 3) administration, one month before (Month 9) and one month after (Month 10) the booster dose of Synflorix™ vaccine
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 156 | 151
IU/mL
  Anti-D, Month 3 (N=154, 151) | 1.791 [1.503 to 2.133] | 3.123 [2.621 to 3.723]
  Anti-D, Month 9 (N= 154, 148) | 0.326 [0.275 to 0.386] | 0.725 [0.622 to 0.846]
  Anti-D, Month 10 (N= 156, 148) | 5.423 [4.815 to 6.108] | 8.262 [7.339 to 9.301]
  Anti-T, Month 3 (N=154, 151) | 2.504 [2.17 to 2.89] | 4.602 [4.062 to 5.213]
  Anti-T, Month 9 (N= 153, 149) | 0.565 [0.487 to 0.656] | 1.191 [1.055 to 1.344]
  Anti-T, Month 10 (N= 156, 148) | 7.678 [6.997 to 8.425] | 9.597 [8.749 to 10.526]

7. Secondary Outcome: Antibody Concentrations Against Polyribosyl Ribitol Phosphate (Anti-PRP)
Description: Concentrations of antibodies are presented as geometric mean concentrations, expressed as micrograms per milliliter (μg/mL). Seroprotection status was defined as anti-polyribosyl ribitol phosphate (Anti-PRP) antibody concentrations greater than or equal to (≥) the cut-off values of 0.15 μg/mL and ≥ 1.0 μg/mL. This outcome concerns results for the Primary and Booster Phases of the study.
Time Frame: One month post-dose 2 (Month 3) administration, one month before (Month 9) and one month after (Month 10) booster dose of Synflorix™ vaccine
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 155 | 148
μg/mL
  Anti-PRP, Month 3 (N=146, 147) | 1.179 [0.893 to 1.556] | 2.186 [1.648 to 2.9]
  Anti-PRP, Month 9 (N=150, 148) | 0.431 [0.349 to 0.532] | 0.777 [0.613 to 0.984]
  Anti-PRP, Month 10 (N=155, 147) | 16.943 [13.485 to 21.287] | 21.654 [17.263 to 27.161]

8. Secondary Outcome: Antibody Concentrations Against Pertussis Toxoid (Anti-PT), Filamentous Haemagglutinin (Anti-FHA) and Pertactin (Anti-PRN)
Description: Concentrations of antibodies are presented as geometric mean concentrations, expressed as enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL). Seropositivity status was defined as anti-pertussis toxoid (Anti-PT), anti-filamentous haemagglutinin (Anti-FHA) and anti-pertactin (Anti-PRN) antibody concentrations greater than or equal to (≥) the cut-off value of 5 EL.U/mL. This outcome concerns results for the Primary and Booster Phases of the study.
Time Frame: One month post-dose 2 (Month 3) administration, one month before (Month 9) and after (Month 10) the booster dose of Synflorix™ vaccine
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 150 | 147
EL.U/mL
  Anti-PT, Month 3 (N=145, 144) | 36.1 [32.9 to 39.6] | 33.8 [30.2 to 37.9]
  Anti-PT, Month 9 (N=144, 145) | 9.8 [8.7 to 11.1] | 10.2 [8.9 to 11.7]
  Anti-PT, Month 10 (N=149, 145) | 78.2 [70.5 to 86.8] | 65.5 [58.7 to 73.1]
  Anti-FHA, Month 3 (N=145, 144) | 166.7 [150.1 to 185.2] | 142.2 [125.6 to 161.1]
  Anti-FHA, Month 9 (N=144, 145) | 46.6 [41.3 to 52.6] | 46.9 [41.1 to 53.6]
  Anti-FHA, Month 10 (N=149, 144) | 360.3 [323.7 to 401] | 276.6 [249.4 to 306.7]
  Anti-PRN , Month 3 (N=145, 144) | 83.9 [69.6 to 101.1] | 89 [74.1 to 106.8]
  Anti-PRN, Month 9 (N=144, 145) | 13.7 [11.2 to 16.6] | 18 [14.8 to 21.8]
  Anti-PRN, Month 10 (N=150, 147) | 275.5 [235.9 to 321.7] | 209.3 [181.8 to 241]

9. Secondary Outcome: Antibody Concentrations Against Hepatitis B Surface Antigen (Anti-HBs)
Description: Concentrations of antibodies are presented as geometric mean concentrations, expressed as milli international units per milliliter (mIU/mL). Seroprotection status was defined as anti-hepatitis B surface antigen (anti-HBs) antibody concentrations greater than or equal to (≥) the cut-off value of 10 mIU/mL. This outcome concerns results for the Primary and Booster Phases of the study and included only the subset of subjects who received Infanrix Hexa™ as the co-administered vaccine.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 40 | 46
mIU/mL
  Anti-HBs, Month 3 (N=37, 38) | 293.7 [195.9 to 440.5] | 478.6 [294.8 to 776.9]
  Anti-HBs, Month 9 (N=40, 46) | 84.3 [55.4 to 128.2] | 156.6 [106.4 to 230.4]
  Anti-HBs, Month 10 (N=27, 28) | 1892.3 [1012.2 to 3537.6] | 2922.4 [2010.4 to 4248.1]

10. Secondary Outcome: Antibody Titers Against Polio Type 1, 2 and 3 (Anti-polio 1, 2 and 3)
Description: Titers of antibodies are presented as geometric mean titers. Seroprotection status was defined as anti-polio types 1, 2 and 3 (Anti-polio 1, 2 and 3) antibody titers greater than or equal to (≥) the value of 8. This outcome concerns results for the Primary and Booster Phases of the study and included only the subset of subjects who received Infanrix Hexa™ as the co-administered vaccine.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 50 | 59
Titers
  Anti-Polio 1, Month 3 (N=47, 57) | 88.5 [56.3 to 139.1] | 99.1 [63.4 to 154.8]
  Anti-Polio 1, Month 9 (N=45, 39) | 24.6 [15.6 to 38.8] | 14.4 [8.9 to 23.1]
  Anti-Polio 1, Month 10 (N=20, 15) | 1006.4 [541.8 to 1869.4] | 645 [399.4 to 1041.7]
  Anti-Polio 2, Month 3 (N=47, 59) | 57.7 [36.8 to 90.6] | 40.5 [25 to 65.6]
  Anti-Polio 2, Month 9 (N=44, 40) | 14.9 [10.7 to 20.9] | 10.9 [7.2 to 16.4]
  Anti-Polio 2, Month 10 (N=17, 14) | 522.4 [235.7 to 1157.7] | 512.2 [186.4 to 1407.7]
  Anti-Polio 3, Month 3 (N=50, 57) | 165.6 [109.3 to 250.8] | 161 [98.7 to 262.8]
  Anti-Polio 3, Month 9 (N=44, 38) | 15.1 [9.8 to 23.2] | 14.7 [9 to 24.1]
  Anti-Polio 3, Month 10 (N=5, 11) | 1910.8 [257.4 to 14185.3] | 961.4 [388.3 to 2380.6]

11. Secondary Outcome: Number of Subjects With Booster Vaccine Response to Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: Booster vaccine response to pertussis toxoid (PT), filamentous haemagglutinin (FHA) and pertactin (PRN), defined as the appearance of antibodies in subjects who were seronegative (Pre-booster status S-) (i.e., with antibody concentrations < 5 EL.U/mL) just before booster dose, and at least two-fold increase of pre-vaccination antibody concentrations in those who were seropositive (Pre-booster status S+) (i.e., with antibody concentrations ≥ 5 EL.U/mL) just before booster dose.
Time Frame: One month after (Month 9) the administration of the booster dose of Synflorix™ vaccine
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 137 | 142
Subjects
  Anti-PT, Pre-booster status S- (N=20, 23) | 20 | 23
  Anti-PT, Pre-booster status S+ (N=117, 117) | 115 | 114
  Anti-PT, Pre-booster status Total (N=137, 140) | 135 | 137
  Anti-FHA, Pre-booster status S- (N=0, 1) | 0 | 1
  Anti-FHA, Pre-booster status S+ (N=137, 138) | 132 | 129
  Anti-FHA, Pre-booster status Total (N=137, 139) | 132 | 130
  Anti-PRN, Pre-booster status S- (N=35, 21) | 35 | 21
  Anti-PRN, Pre-booster status S+ (N=102, 121) | 101 | 119
  Anti-PRN, Pre-booster status Total (N=137, 142) | 136 | 140

12. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed local symptoms were pain, redness and swelling. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm). Across doses= across the 2 doses of the Synflorix™ vaccine in the Synflorix I group and across the 3 doses of the Synflorix™ vaccine in the Synflorix II group.
Time Frame: During the 4-day (Days 0-3) period following the primary vaccination (across doses) and during the 4-day (Days 0-3) period following the booster vaccination (post Booster) with the Synflorix™ vaccine
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects (i.e. who had received at least one dose of study vaccine during the primary vaccination course or the booster dose).
Measure: Number; unit: Subjects
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 175 | 176
Subjects
  Any Pain, across doses (N=175; 176) | 92 | 110
  Grade 3 Pain, across doses (N=175; 176) | 14 | 12
  Any Redness, across doses (N=175; 176) | 137 | 135
  Grade 3 Redness, across doses (N=175; 176) | 4 | 6
  Any Swelling, across doses (N=175; 176) | 111 | 105
  Grade 3 Swelling, across doses (N=175; 176) | 20 | 16
  Any Pain, post Booster (N=174, 169) | 103 | 93
  Grade 3 Pain, post Booster (N=174, 169) | 7 | 5
  Any Redness, post Booster (N=174, 169) | 118 | 115
  Grade 3 Redness, post Booster (N=174, 169) | 20 | 20
  Any Swelling, post Booster (N=174, 169) | 97 | 99
  Grade 3 Swelling, post Booster (N=174, 169) | 19 | 15

13. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability/fussiness (Irr./Fuss.), loss of appetite (Loss Appet.) and fever (rectal temperature higher than [≥] 38.0 degrees Celsius [°C]). Any = Occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Related = Occurrence of the specified symptom assessed by the investigators as causally related to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irr./Fuss. = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. Grade 3 Fever = Rectal temperature higher than (>) 40.0°C. Across doses= across the 2 doses of the Synflorix™ vaccine in the Synflorix I group and across the 3 doses of the Synflorix™ vaccine in the Synflorix II group.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Number; unit: Subjects
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 175 | 176
Subjects
  Any Drowsiness, across doses (N=175, 176) | 130 | 130
  Grade 3 Drowsiness, across doses (N=175, 176) | 9 | 4
  Related Drowsiness, across doses (N=175, 176) | 123 | 124
  Any Fever, across doses (N=175, 176) | 108 | 116
  Grade 3 Fever, across doses (N=175, 176) | 0 | 0
  Related Fever, across doses (N=175, 176) | 106 | 108
  Any Irr./Fuss., across doses (N=175, 176) | 149 | 158
  Grade 3 Irr./Fuss., across doses (N=175, 176) | 18 | 28
  Related Irr./Fuss., across doses (N=175, 176) | 142 | 147
  Any Loss Appet., across doses (N=175, 176) | 81 | 88
  Grade 3 Loss Appet., across doses (N=175, 176) | 5 | 1
  Related Loss Appet., across doses (N=175, 176) | 75 | 81
  Any Drowsiness, post Booster (N=174, 169) | 97 | 79
  Grade 3 Drowsiness, post Booster (N=174, 169) | 6 | 2
  Related Drowsiness, post Booster (N=174, 169) | 83 | 71
  Any Fever, post Booster (N=174, 169) | 96 | 78
  Grade 3 Fever, post Booster (N=174, 169) | 1 | 0
  Related Fever, post Booster (N=174, 169) | 84 | 67
  Any Irr./Fuss., post Booster (N=174, 169) | 113 | 104
  Grade 3 Irr./Fuss., post Booster (N=174, 169) | 6 | 2
  Related Irr./Fuss., post Booster (N=174, 169) | 99 | 89
  Any Loss Appet., post Booster (N=174, 169) | 61 | 56
  Grade 3 Loss Appet., post Booster (N=174, 169) | 3 | 0
  Related Loss Appet., post Booster (N=174, 169) | 53 | 43

14. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events
Description: An unsolicited AE was defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For the marketed products administered in the study, this also included failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse of the product. Any = Occurrence of an unsolicited AE, regardless of intensity or relationship to vaccination.
Time Frame: Within the 31-day (Days 0-30) post-primary vaccination period, across doses
Population: as for outcome 12
Measure: Number; unit: Subjects
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 175 | 176
Subjects | 78 | 114

15. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events
Description: as for outcome 14
Time Frame: Within the 31-day (Days 0-30) post booster vaccination period
Population: as for outcome 12
Measure: Number; unit: Subjects
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 174 | 171
Subjects | 63 | 72

16. Secondary Outcome: Number of Subjects With Serious Adverse Events
Description: A SAE was defined as any medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject. AE(s) considered as SAE(s) also included invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalisation, as per the medical or scientific judgement of the physician. Any = Occurrence of a SAE, regardless of relationship to vaccination.
Time Frame: During the primary vaccination period
Population: as for outcome 12
Measure: Number; unit: Subjects
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 175 | 176
Subjects | 5 | 7

17. Secondary Outcome: Number of Subjects With Serious Adverse Events
Description: as for outcome 16
Time Frame: During the booster vaccination period
Population: as for outcome 12
Measure: Number; unit: Subjects
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 174 | 171
Subjects | 2 | 1

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4 days post-primary vaccination (across doses) and post-booster dose. Unsolicited AEs: during 31 days post-primary vaccination (across doses) and post-booster dose. SAEs: during both primary and booster vaccination periods.
Description: Analysis of AEs and SAEs was done on subjects with at least 1 primary vaccination dose. Analysis of solicited symptoms was done on subjects with at least 1 primary dose and with results available. Occurrences (all and "related to the treatment") were not calculated during the analysis and are filled in with "subjects affected" similar information.
Arm/Group | Synflorix I Group | Synflorix II Group
Serious Adverse Events (participants affected / at risk) | 5/175 | 7/176
Other Adverse Events (participants affected / at risk) | 173/175 | 175/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Synflorix I Group (N=175) | Synflorix II Group (N=176)
Asthma (Primary phase) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Febrile convulsion (Booster phase) (Nervous system disorders) | 1/174 | 0/171
Dyspepsia (Primary phase) (Gastrointestinal disorders) | 0 | 1
Dermatitis allergic (Primary phase) (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory syncytial virus infection (Primary phase) (Infections and infestations) | 1 | 1
Bronchopneumonia (Primary phase) (Infections and infestations) | 0 | 1
Gastroenteritis (Primary phase) (Infections and infestations) | 0 | 1
Gastroenteritis viral (Primary phase) (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Primary phase) (Infections and infestations) | 0 | 1
Salmonellosis (Primary phase) (Infections and infestations) | 1 | 0
Tracheitis (Primary phase) (Infections and infestations) | 0 | 1
Urinary tract infection (Primary phase) (Infections and infestations) | 0 | 1
Viral infection (Primary phase) (Infections and infestations) | 1 | 0
Otitis media (Booster phase) (Infections and infestations) | 0/174 | 1/171
Pneumonia (Booster phase) (Infections and infestations) | 1/174 | 0/171
Urinary tract infection (Booster phase) (Infections and infestations) | 1/174 | 0/171
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Synflorix I Group (N=175) | Synflorix II Group (N=176)
Cough (Primary phase) (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Cough (Booster phase) (Respiratory, thoracic and mediastinal disorders) | 6/174 | 11/171
Pain (Primary phase) (General disorders) | 92 | 110
Redness (Primary phase) (General disorders) | 137 | 135
Swelling (Primary phase) (General disorders) | 111 | 105
Pain (Booster phase) (General disorders) | 103/174 | 93/169
Redness (Booster phase) (General disorders) | 118/174 | 115/169
Swelling (Booster phase) (General disorders) | 97/174 | 99/169
Drowsiness (Primary phase) (General disorders) | 130 | 130
Fever- rectal (Primary phase) (General disorders) | 108 | 116
Irritability (Primary phase) (General disorders) | 149 | 158
Loss of appetite (Primary phase) (General disorders) | 81 | 88
Drowsiness (Booster phase) (General disorders) | 97/174 | 79/169
Fever- rectal (Booster phase) (General disorders) | 96/174 | 78/169
Irritability (Booster phase) (General disorders) | 113/174 | 104/169
Loss of appetite (Booster phase) (General disorders) | 61/174 | 56/169
Pyrexia (Primary phase) (General disorders) | 12 | 12
Pyrexia (Booster phase) (General disorders) | 8/174 | 10/171
Diarrhoea (Gastrointestinal disorders) | 11 | 8
Vomiting (Gastrointestinal disorders) | 4 | 10
Nasopharyngitis (Primary phase) (Infections and infestations) | 26 | 46
Nasopharyngitis (Booster phase) (Infections and infestations) | 16/174 | 20/171
Otitis media (Booster phase) (Infections and infestations) | 9/174 | 7/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.